CLINICAL TRIAL: NCT05834517
Title: ''Efficacy of Locally Delivered Hyaluronic Acid Gel as an Adjunctive to Non-Surgical Management of Stage II or Stage III Periodontitis
Brief Title: ''Efficacy of Locally Delivered Hyaluronic Acid Gel as an Adjunctive to Non-Surgical Management of Periodontitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ehab Haider Hassan El-emam (Other)
Responsible Party: Sponsor-Investigator, Ehab Haider Hassan El-emam, ehab haider hassan elemam, Ain Shams University
Organization: Ain Shams University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FDASU-RECD125091
Record Dates: First submitted 2023-04-17; First posted 2023-04-28 (Actual); Last update posted 2023-04-28 (Actual); Status verified 2023-04

CONDITIONS: Periodontitis
MeSH Terms: conditions — Periodontitis | interventions — Hyaluronic Acid

STUDY DESIGN:
Intervention Model Description: topical application of hyaluronic acid in patients with periodontitis 1 day after scaling
Who Masked: Outcomes Assessor
Masking Description: The eligible participants will be randomly allocated for one of the two groups; test and control group using computer generated random tables.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- hyaluronic acid/ scaling (Experimental): topical application of hyaluronic acid after scaling by 1 day
  Interventions: Drug: Hyaluronic acid; Procedure: non surgical periodontal therapy
- scaling (Experimental): scaling only
  Interventions: Procedure: non surgical periodontal therapy

INTERVENTIONS:
Drug: Hyaluronic acid — Hyaluronic Acid (HA) is an addition to the local chemotherapeutic agents. Hyaluronic acid was discovered by Meyer and Palmer. HA is widely found in the extracellular matrix and it plays an essential role in controlling cell behavior including random motility, metabolic reactions, chemotaxis, proliferation and invasion. HA is released by many cells including fibroblasts
  Other Names: hyaluronan
  Arms: hyaluronic acid/ scaling
Procedure: non surgical periodontal therapy — NSPT, with or without adjunctive therapies, is an effective treatment for periodontitis. It reduces PD and results in formation of some new attachment; however, it also has several limitations, and surgical therapy might be required to control inflammation and optimize outcomes. When used for non-surgical scaling and root planing, periodontal curettes can reach a mean PD of up to approximately 5.5 mm. The mean PD in which a plaque-free and calculus-free surface can be established is <4 mm

SUMMARY:
Hyaluronic Acid (HA) is an addition to the local chemotherapeutic agents. Hyaluronic acid was discovered by Meyer and Palmer. HA is widely found in the extracellular matrix and it plays an essential role in controlling cell behavior including random motility, metabolic reactions, chemotaxis, proliferation and invasion. HA is released by many cells including fibroblasts (Dahiya et al., 2013).

Hyaluronic acid can be found in the skin, eyes and the periodontium. In addition, it appears in body fluids like serum, gingival crevicular fluid and saliva. Hyaluronic acid is created in the periodontium by HA synthase enzyme present in numerous cells like fibroblast and cementoblast (Fraser et al., 1997).

There is evidence that hyaluronic acid is bacteriostatic, fungostatic, anti-inflammatory, osteoconduvtive and pro-angiogenic. These dissimilar properties illustrate the ability of hyaluronic acid to be an ideal material for wound healing (Carlson et al., 2004).

DETAILED DESCRIPTION:
Periodontitis is a chronic multifactorial inflammatory disease, associated with the dental plaque biofilms, its distinct feature is destruction of the tooth supporting apparatus. Its main features include: damage of the periodontal tissue, that's manifested by clinical attachment loss, alveolar bone loss, periodontal pocketing and bleeding gum (Armitage, 1999).

A new periodontitis classification scheme has been approved, in which forms of the disease previously known as "chronic" or "aggressive" are now gathered under a single term ("periodontitis") and are more characterized based on a multi-dimensional staging and grading system. Staging is basically reliant on the severity of disease as well as on the difficulty of disease management, on the other hand , grading offers additional information about biological aspects of the disease including a history-based analysis of the rate of periodontitis progression; risk assessment for further progression and analysis of likely poor outcomes of treatment (Caton et al., 2018; Papapanou et al., 2018).

Host-Microbial interaction is having a huge effect on the nature of periodontal disease progression. The microbial biofilm elicits the host to release inflammatory mediators that have a negative effect on the connective tissues. The biofilm or dental plaque is required but not enough to induce periodontitis, since it is the host inflammatory response to this microbial challenge that eventually can be the reason for destruction of the periodontium (Haffajee and Socransky, 1994; Page , 1997; Darveau, 2010).

Physical removal of dental plaque through debridement and/or using antimicrobial agents is the most prevalent management of periodontitis. Initially, scaling and root planing (SRP) is done with the means of hand or ultrasonic instruments to debride the root surface, allowing the development of a long junctional epithelium. Clinically, in case of lack of accessibility like extensive tissue loss, deep periodontal pocket and furcation involvement make it unclear to determine the efficacy of the debridement (Lindhe, 1985).

The use systemic antibiotics (ABs) can contribute in treatment goals without surgical treatment. However, their usage is limited to particular patients for those who have previously two courses of SRP with no improvement in periodontal pocket depth. Additionally, the side effects and rise in AB resistance over time have reduced the number of cases managed in this way (Walters et al., 2015).

Local antimicrobial therapy includes the direct placement of an antimicrobial agent into sub gingival sites, limiting the effect of the agent on non-oral body sites. The main goal in using an intra-pocket device for the delivery of an antibacterial agent is maintenance of therapeutic levels of the drug for the required period of time. This method has direct influence on the pathogens, without any damage to the tissues (Garg, 2015).

The first local drug delivery system in periodontal treatment was ActiciteTM. The first non resorbable system. Although quite effective, the delivery of this system in the periodontal pockets required extra skills and another visit to the dentist in order to be removed. The drawbacks of the non-resorbable systems headed to the advance of resorbable systems for antimicrobial delivery like ATRIDOXTM, gel containing 10 % doxycyline hyclate. Progresses in the formulation of local delivery systems lead to the manufacture of ARESTINTM, sustained release product consist of minocycline (Krayer et al., 2010).

Local delivery antibiotics that are commercially available as controlled release devices had many disadvantages including limited spectrum of antimicrobial activity in some periodontal polymicrobial infections, risk of generating antimicrobial resistance and massive acquisition cost (Sltos , 2002).

The most extensive used and studied antiseptic in oral diseases is chlorhexidine. Chlorhexidine displays high affinity towards bacteria .The highest advantages of chlorhexidine application after SRP or surgical periodontal treatment include better-quality in wound healing and general plaque control (Horz & Conrads, 2007). However, even with the advantages, the application may end with staining of the teeth, taste disturbances and increase of calculus formation (Zanatta et al., 2010).

Hyaluronic Acid (HA) is an addition to the local chemotherapeutic agents. Hyaluronic acid was discovered by Meyer and Palmer. HA is widely found in the extracellular matrix and it plays an essential role in controlling cell behavior including random motility, metabolic reactions, chemotaxis, proliferation and invasion. HA is released by many cells including fibroblasts (Dahiya et al., 2013).

Hyaluronic acid can be found in the skin, eyes and the periodontium. In addition, it appears in body fluids like serum, gingival crevicular fluid and saliva. Hyaluronic acid is created in the periodontium by HA synthase enzyme present in numerous cells like fibroblast and cementoblast (Fraser et al., 1997).

There is evidence that hyaluronic acid is bacteriostatic, fungostatic, anti-inflammatory, osteoconduvtive and pro-angiogenic. These dissimilar properties illustrate the ability of hyaluronic acid to be an ideal material for wound healing (Carlson et al., 2004).

The anti-inflammatory action of hyaluronic acid is related to the role of exogenous Hyaluronan as a scavenger by draining metaloprotinases, prostaglandins and other bio-active molecules (Laurant et al., 1995). Moreover, hyaluronic acid is anti-edematous due to its osmotic activity. The high concentration of medium and lower molecular weight hyaluronic acid has a possible bacteriostatic role especially on aggregatibacter actinomyecetemcomitans and staph aureus strains which are usually found in periodontal wounds (Pirnazar et al., 1999).

In patients with chronic periodontitis, the adjunctive application of hyaluronic acid to non -surgical periodontal treatment including (scaling and root planning) results in much higher clinical improvement including probing depth and bleeding on probing (Bertl, 2015).

A clinical trial by (Yi Xu et al ., 2004) used HA gel as an adjunctive to scaling and root planning in treatment of chronic periodontitis , regarding the clinical parameters and microbiological analysis had revealed that HA gel has an essential role in improvement of all clinical parameters but in contrary, microbiological analysis using conventional PCR revealed that hyaluronic acid has no effect on the bacteria .

Based on the previously mentioned properties hyaluronic acid, We hypothesized that hyaluronic acid has a major role to be used as an adjunctive to non-surgical treatment in periodontitis patients.

ELIGIBILITY:
Inclusion Criteria:

.Patients have to be free from any systemic disease as proven by Burket's oral medicine health history questionnaire (Glik et al., 2008).

.Both genders aged 20-55.

. Periodontitis (Stage II or stage III) Patients; (3-6 mm CAL ,pocket depth ≤7 mm, mostly horizontal 15%-33% bone loss as assessed by preoperative radiographs with no tooth loss due to periodontitis) (Tonetti et al., 2017).

Exclusion Criteria:

* Pregnant lactating females
* Smoking
* Patients who can't be committed to oral hygiene instructions
* History of periodontal surgery or antimicrobial therapy for at least 4 months.

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2022-05-02 (Actual); Primary Completion 2022-12-05 (Actual); Study Completion 2022-12-10 (Actual)

PRIMARY OUTCOMES:
clinical score | 3 months
  1-Plaque index (PI) 2. Sulcus bleeding index (BI) 3-Probing depth (PD) 4-Clinical attachment loss level (CAL)

SECONDARY OUTCOMES:
analyzing quantitative changes of pathogenic periodontal bacteria as a secondary objectives. | 1 month
  using real time PCR for analyzing the bacterial loads of 1. Porphyromonus gingivalis 2. Aggregatibacter Actinomycetumomitans

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No